CLINICAL TRIAL: NCT07041762
Title: Analgesic Efficacy of Rhomboid Intercostal Block With Sub-Serratus Plane Block Versus Erector Spinae Block in Breast Cancer Surgery
Brief Title: Rhomboid Intercostal Block With Sub-Serratus Plane Block Versus Erector Spinae Block
Acronym: RISS-ESPB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sayed Mahmoud Abed, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCI-CAIRO-RISS-ESPB-2025
Record Dates: First submitted 2025-06-10; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Patients
Keywords: erector spinae block

STUDY DESIGN:
Intervention Model Description: double blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind design: Participants, anesthesia providers, investigators, and outcome assessors will be blinded to group allocation. Group assignments will be concealed using opaque sealed envelopes, and blocks will be performed by anesthesiologists not involved in intraoperative care or postoperative evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhomboid Intercostal Block with Sub-Serratus Plane Block (Experimental): Participants in this group will receive ultrasound-guided Rhomboid Intercostal Block (20 mL of 0.25% bupivacaine between rhomboid major and intercostal space) followed by Sub-Serratus Plane Block (20 mL of 0.25% bupivacaine between serratus anterior and ribs) 30-45 minutes before general anesthesia for Modified Radical Mastectomy.
  Interventions: Procedure: Rhomboid Intercostal Block with Sub-Serratus Plane Block
- Erector Spinae Plane Block (Active Comparator): Participants in this group will receive an ultrasound-guided Erector Spinae Plane Block with 30 mL of 0.25% bupivacaine injected into the paraspinal plane at the T4-T5 level, 30-45 minutes prior to general anesthesia for Modified Radical Mastectomy.
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Rhomboid Intercostal Block with Sub-Serratus Plane Block — Ultrasound-guided regional anesthesia combining two injections:
  Rhomboid Intercostal Block (20 mL of 0.25% bupivacaine injected between rhomboid major and intercostal space)
  Sub-Serratus Plane Block (20 mL of 0.25% bupivacaine injected between serratus anterior and ribs).
  Both performed 30-45 minutes before Modified Radical Mastectomy under general anesthesia.
  Arms: Rhomboid Intercostal Block with Sub-Serratus Plane Block
Procedure: Erector Spinae Plane Block — Ultrasound-guided regional block with 30 mL of 0.25% bupivacaine injected into the paraspinal plane at the T4-T5 level, between the erector spinae muscle and the transverse processes.
  Performed 30-45 minutes prior to general anesthesia for Modified Radical Mastectomy.
  Arms: Erector Spinae Plane Block

SUMMARY:
This study compares two nerve block techniques-Rhomboid Intercostal with Sub-Serratus Plane Block versus Erector Spinae Plane Block-for pain relief after breast cancer surgery. It aims to determine which method provides better postoperative pain control, reduces opioid use, and improves recovery in patients undergoing modified radical mastectomy at the National Cancer Institute, Cairo University.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the analgesic efficacy of two ultrasound-guided regional anesthesia techniques-Rhomboid Intercostal Block with Sub-Serratus Plane Block (RIB + SSP) and Erector Spinae Plane Block (ESB)-in patients undergoing Modified Radical Mastectomy (MRM) for breast cancer. Eighty female patients aged 18-65 years with ASA physical status II or III will be enrolled and randomly assigned to receive either RIB + SSP or ESB prior to surgery. Both blocks will be performed under ultrasound guidance 30-45 minutes before induction of general anesthesia.

The primary outcomes are postoperative pain scores measured using the Visual Analog Scale (VAS) and total opioid consumption in the first 24 hours after surgery. Secondary outcomes include intraoperative and postoperative hemodynamic parameters, time to first analgesic request, total intraoperative opioid use, recovery time, patient satisfaction, and incidence of adverse effects such as nausea and vomiting.

The study will be conducted at the National Cancer Institute - Cairo University from June 2025 to June 2026. Ethical approval will be obtained, and written informed consent will be collected. This study aims to identify the more effective and safer regional technique to improve postoperative recovery and reduce opioid dependence in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients undergoing Modified Radical Mastectomy (MRM)

ASA physical status II or III

Age between 18 and 65 years

Body Mass Index (BMI) > 20 kg/m² and < 35 kg/m²

Exclusion Criteria:

* Patient refusal

ASA physical status IV

Age <18 years or >65 years

BMI < 20 kg/m² or > 35 kg/m²

Known allergy or contraindication to local anesthetics or opioids

History of psychological disorders or chronic pain

Contraindications to regional anesthesia (e.g., coagulopathy, local infection, peripheral neuropathy)

Severe respiratory, cardiac, hepatic, or renal disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Scores | First 24 hours postoperatively
  Postoperative pain will be assessed using the Visual Analog Scale (VAS) both at rest (static) and during movement (dynamic). Assessments will be conducted at 2, 6, 12, and 24 hours following surgery. The VAS is a 10-centimeter scale, where 0 indicates "no pain" and 10 indicates the "worst imaginable pain." Unit of Measure: VAS score (0-10)
Total Opioid Consumption | First 24 hours postoperatively
  The total amount of opioid analgesics administered within the first 24 postoperative hours will be recorded for each patient. All opioid dosages will be converted to intravenous morphine equivalents for standardization.
  Unit of Measure: Milligrams of intravenous morphine equivalents (mg)

CONTACTS AND LOCATIONS:
Overall Officials: Sayed Mahmoud M Abed, MD, Principal Investigator — National Cancer Institute - Cairo University
Locations (1):
- National Cancer Institute - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to institutional policies regarding data confidentiality and privacy. Additionally, there is no established infrastructure for secure data sharing or monitoring of secondary data use at this time.

REFERENCES:
- See also: Rhomboid intercostal block combined with sub-serratus plane block versus rhomboid intercostal block for postoperative analgesia after video-assisted thoracoscopic surgery: a prospective randomized-controlled trial — https://pubmed.ncbi.nlm.nih.gov/33632189/
- See also: Rhomboid Intercostal and Subserratus Plane Block: A Cadaveric and Clinical Evaluation — https://rapm.bmj.com/content/43/7/745